CLINICAL TRIAL: NCT04341324
Title: Prospective Study of the Effect of Androgen Deprivation Therapy (ADT) in Male Patients Suffered Prostate Cancer in Chinese Population
Brief Title: Effect of ADT in Chinese Male With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRE 2010.577-T
Record Dates: First submitted 2020-04-02; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for fasting lipid, sugar, hsCRP and other hormones (about 15cc) will be assessed in each study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active arm: Subjects received hormonal therapy: Study subject inclusion criteria
  1. Male patients 18 years or older
  2. Adenocarcinoma of the prostate either histologically or cytologically confirmed
  3. Decided to be put on ADT -bilateral orchidectomy or luteinizing hormone-releasing hormone (LHRH) agonist or LHRH antagonist, with or without additional antiandrogen
  4. After ADT performed, serum testosterone level should reach castrated level, i.e. < 50 ng/dL after 6 weeks of treatment
  5. Able to consent for the participate in the study
  Interventions: Other: It is an observational study.
- Control arm: Subjects do not plan to receive hormonal therapy: Control subject:
  1. Male patients 18 years or older
  2. Adenocarcinoma of the prostate either histologically or cytologically confirmed
  3. Able to consent for the participate in the study

INTERVENTIONS:
Other: It is an observational study.
  Groups: Active arm: Subjects received hormonal therapy

SUMMARY:
Many prostate cancer patients required the use of androgen deprivation therapy (ADT) for the control of disease.

In this study, the investigators aim at assessing the different in various parameters between PCa patients received ADT and those without ADT.

60 patients diagnosed with PCa and planned for hormonal therapy will be recruited for study (active arm) and 30 PCa patients that do not planned to receive hormonal therapy (based on the clinical assessment by the investigators) will be recruited as control arm.

After written consent obtained from study subject, a series of investigation will be arranged to assess the following aspect of the subjects before the commenced of ADT:

* General condition - symptoms, general health,
* Body composition - BMI and body composition
* Mental state assessment by Mini-Mental State Examination (MMSE)
* Blood for fasting lipid, sugar, hsCRP and other hormones (about 15cc)
* Cardiovascular status - BP, Ankle-brachial index (ABI), Arterial stiffness, ECG,
* Bone status - bone mineral density by dual-energy X-ray absorptiometry (DEXA) scan

The assessment of general condition, body composition, blood parameter and cardiovascular status will be performed every 26weeks +/- 1 weeks for two years. Bone density measurement will be performed every 52 weeks +/- 2 weeks.

Appropriate medical referral will be made if subject was found to have abnormal metabolic or cardiovascular parameters.

DETAILED DESCRIPTION:
The prostate gland is a clinically important male accessory sex gland and vital for its production of semen. Prostate cancer (PCa) is now ranked 4th in annual incidence of male cancer and ranked 8th for cancer-related death in men in Hong Kong which accounts for about 6.2 deaths per 100,000 persons. Its incidence is rising rapidly, almost tripled in the past 10 years. As the elderly population continues to increase, the impact of PCa on the men's health and also the burden on health care system will continue to rise.

Despite the improvement in awareness of the disease and also increasing use of serum prostate specific antigen, many patients still presented at a late stage that beyond cure by local therapy. Together with those patients suffered recurrent disease after local therapy, many PCa patients required the use of androgen deprivation therapy (ADT) for the control of disease.

However, unlike other malignancy, PCa is characterized by its slow progression nature and even for metastatic disease the 5-year survival is upto 20%. Therefore, while ADT can provide effective control of disease, there are increasing evidences suggesting that it can also result in many adverse effects in the patients, and these effects are particular important due to the long survival of these patients. From the western literature, the adverse effects can be quite diverse. Classical side effects after ADT include mood changes, hot flushes, change in cognitive function, loss of libido, erectile dysfunction, osteoporosis and pathological fracture. Also there are more and more evidences showed ADT will also altered the metabolic and cardiovascular status of the patients and resulted in increase in insulin resistance and increase in risk of cardiovascular related mortality.

Traditionally, in order to achieve a complete control of PCa, ADT is given in a continue manner, either in the form of bilateral orchidectomy or regular luteinizing hormone releasing hormone injection. However, in order to balance the benefit and potential of long-term complication, intermittent hormonal therapy (IHT) become increasing common to be used in patients suffered PCa, in particular those with low tumour volume and low-grade disease. However, formal comparison of the benefit, in term of side effect reduction, for IHT compare to traditional continue-hormonal suppression is still lacking.

Unfortunately information regarding the side effects of ADT in Chinese population is lacking. However, there are some evidences from female menopause related studies that there may be some differences in the presentation and prevalence of sex hormone deprivation in difference racial groups. Therefore, there is a need to have more information on the adverse effect profiles related to ADT (both complete and IHT) in Chinese population.

ELIGIBILITY:
For those received hormonal therapy will be recruited for study (active arm) Study subject inclusion criteria

1. Male patients 18 years or older
2. Adenocarcinoma of the prostate either histologically or cytologically confirmed
3. Decided to be put on ADT -bilateral orchidectomy or LHRH agonist or LHRH antagonist, with or without additional antiandrogen
4. After ADT performed, serum testosterone level should reach castrated level, i.e. < 50 ng/dL after 6 weeks of treatment
5. Able to consent for the participate in the study

For those do not plan to receive hormonal therapy (based on the clinical assessment by the investigators) will be recruited as control arm

Control subject:

1. Male patients 18 years or older
2. Adenocarcinoma of the prostate either histologically or cytologically confirmed
3. Able to consent for the participate in the study

Exclusion Criteria:

1. Patient did not able to provide consent or comply with the follow-up arrangement
2. Patient with life expectancy of less than 2 years - based on clinical judgement

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only mole can develop prostate cancer
Study Population: 60 patients diagnosed with PCa will be recruited for the study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-07-14 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline cardiovascular risk at 24 months | At baseline and month-24
  Measured by Framingham risk score (Estimation of 10-year Cardiovascular Disease Risk in percentage)

SECONDARY OUTCOMES:
Change from Baseline total cholesterol at 24 months | At baseline and month-24
  Measured by total cholesterol blood test
Change from Baseline low density lipoprotein at 24 months | At baseline and month-24
  Measured by low density lipoprotein blood test
Change from Baseline high-density lipoprotein at 24 months | At baseline and month-24
  Measured by high-density lipoprotein blood test
Change from Baseline triglyceride at 24 months | At baseline and month-24
  Measured by triglyceride blood test
Change from Baseline body mass index (BMI) at 24 months | At baseline and month-24
  Weight and height will be combined to report BMI in kg/m^2
Change from Baseline body composition at 24 months | At baseline and month-24
  Measured by percentage of body fat
Change from Baseline mental state at 24 months | At baseline and month-24
  Measured by the General Practitioner assessment of Cognition (GPCOG). Range of total score: 0-9, higher score mean less cognitive impairment (ie. better outcome).
Change from Baseline vascular arterial stiffness at 24 months | At baseline and month-24
  Vascular arterial stiffness measured by Pulse Wave Velocity (m/s) using non-invasive vascular screening device
Change from Baseline ankle brachial index (ABI) at 24 months | At baseline and month-24
  ABI (ratio of the blood pressure at the ankle to the blood pressure in the upper arm) measured by using non-invasive vascular screening device
Compare cardiovascular events | At month-24
  Measured by the cardiovascular adverse event rate
Change from Baseline bone mineral density at 24 months | At baseline and month-24
  Bone mineral density measured by using bone density scanning device
Compare skeletal related events | At month-24
  Measured by the fracture rate

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong

REFERENCES:
- [Background] Beauchet O. Testosterone and cognitive function: current clinical evidence of a relationship. Eur J Endocrinol. 2006 Dec;155(6):773-81. doi: 10.1530/eje.1.02306. PMID 17132744
- [Background] Fang LC, Merrick GS, Wallner KE. Androgen deprivation therapy: a survival benefit or detriment in men with high-risk prostate cancer? Oncology (Williston Park). 2010 Aug;24(9):790-6, 798. PMID 20923031
- [Background] Lattouf JB, Saad F. Bone complications of androgen deprivation therapy: screening, prevention, and treatment. Curr Opin Urol. 2010 May;20(3):247-52. doi: 10.1097/MOU.0b013e32833835be. PMID 20224416
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. Circulation. 2010 Feb 16;121(6):833-40. doi: 10.1161/CIRCULATIONAHA.109.192695. Epub 2010 Feb 1. No abstract available. PMID 20124128
- [Background] Rampp T, Tan L, Zhang L, Sun ZJ, Klose P, Musial F, Dobos GJ. Menopause in German and Chinese women--an analysis of symptoms, TCM-diagnosis and hormone status. Chin J Integr Med. 2008 Sep;14(3):194-6. doi: 10.1007/s11655-008-0194-1. Epub 2008 Oct 14. PMID 18853115
- [Background] Saylor PJ, Smith MR. Metabolic complications of androgen deprivation therapy for prostate cancer. J Urol. 2009 May;181(5):1998-2006; discussion 2007-8. doi: 10.1016/j.juro.2009.01.047. Epub 2009 Mar 14. PMID 19286225
- [Background] Smith MR. Treatment-related diabetes and cardiovascular disease in prostate cancer survivors. Ann Oncol. 2008 Sep;19 Suppl 7(Suppl 7):vii86-90. doi: 10.1093/annonc/mdn458. No abstract available. PMID 18790986
- [Background] Taylor LG, Canfield SE, Du XL. Review of major adverse effects of androgen-deprivation therapy in men with prostate cancer. Cancer. 2009 Jun 1;115(11):2388-99. doi: 10.1002/cncr.24283. PMID 19399748